CLINICAL TRIAL: NCT01942863
Title: Effect of Water Exchange Method on Intubation Depth and Diagnostic Yield in Patients Undergoing Single-balloon Enteroscopy: a Prospective, Randomized, Controlled, Patient-blind Trial.
Brief Title: Effect of Water Exchange Method on Single-balloon Enteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 20131106-6
Record Dates: First submitted 2013-08-02; First posted 2013-09-16 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Single Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water exchange single balloon enteroscopy (Experimental)
  Interventions: Procedure: water exchange single balloon enteroscopy; Other: Procedural Requirements
- CO2 insufflation single balloon enteroscopy (Active Comparator)
  Interventions: Procedure: CO2 insufflation single balloon enteroscopy; Other: Procedural Requirements

INTERVENTIONS:
Procedure: water exchange single balloon enteroscopy — Oral enteroscopy was performed first, followed by the anal route on the same day or later. For oral route, SBE was first advanced beyond Treitz ligation with CO2 insufflation. Then the water exchange method was used for further insertion. Briefly, residual air in the lumen was suctioned, and 37°C water was infused with a peristaltic pump through the biopsy channel to obtain lumen visualization. Turbid luminal water due to residual feces was suctioned and replaced by clean water until the small bowel lumen was clearly visualized again. Thus, infused water was removed predominantly during the insertion phase. The total volume of water was not restricted. For anal route, water exchange or CO2 insufflation method was used from the beginning of insertion respectively.
  Arms: water exchange single balloon enteroscopy
Procedure: CO2 insufflation single balloon enteroscopy — Conventional enteroscopy was performed as CO2 insufflated during insertion. Oral enteroscopy was performed first, followed by the anal route on the same day or later.
  Arms: CO2 insufflation single balloon enteroscopy
Other: Procedural Requirements — SBE was advanced as deeply as possible and complete small bowel visualization was attempted. When the following conditions were met, tattooing at the deepest position with India ink was performed and the endoscope was withdrawn: no further endoscopic advancement could be achieved, detection of a significant lesion and no other lesions suspected, severe stricture, obvious sedation and SBE-related adverse events happened which required termination of further intubation.

SUMMARY:
Enteroscopy, including double balloon enteroscopy (DBE), single balloon enteroscopy (SBE) and spiral enteroscopy (SE) currently, have shown good performances in small bowel diagnostics and seem to be useful in the clinical routine. However, enteroscopy is a time-consuming procedure. During common practice, large volumes of air need to be insufflated for good visualization. It leads to significant distention of the small bowel during the examination, which makes further intubation more technically challenging because of the formation of distended bowel loops and acute angulations and limits the maximal intubation length. According to the published data, the oral insertion depth of different kinds of enteroscopy is limited to approximately 240 cm. The total examination rate range form 18% to 86% for DBE and 0% to 11% for SBE.

It is thought that the intubation depth in small bowel determines the diagnostic yield and the following treatment. The deeper the enteroscopy is advanced into the small bowel, the more lesions may be found and treated. In order to improve the intubation depth of balloon enteroscopy, several methods, such as carbon dioxide insufflation and decompression side tube-equipped device, have been tried and showed positive effects. CO2 insufflation could also reduce severe pain during DBE and residual gas retention after the procedure because of rapid absorption. However, it is not known how much CO2 insufflation can decrease the distention of small bowel and the formation of bowel loops.

Recently, the use of water infusion in lieu of air insufflation has been shown to facilitate completion of colonoscopy, even in potentially difficult patients with prior abdominal or pelvic surgery. Water exchange method obviates excessive lengthening of the colon and the formation of acute angulation, which may cause less pain and easier intubation during scope insertion. Recently, water exchange method was also tried in two patients undergoing SBE via antegrade route in our center. Distal ileum 8cm near to ICV and the cecum was reached respectively (unpublished data), indicating water exchange be a useful method for deep intubation of SBE.

Here a prospective, randomized, controlled trial was designed to investigate whether, compared with CO2 insufflation method, water exchange method could increase the intubation depth and diagnostic yield in patients undergoing SBE.

ELIGIBILITY:
Inclusion Criteria:

* Suspected small-bowel disease

Exclusion Criteria:

* Prior small-bowel surgery
* Total examination of small bowel not planned when image modalities showed
* lesions obviously located on duodenum, proximal jejunum or distal ileum
* High-risk esophageal varices
* Pregnancy or lactation
* Inability to tolerate sedation or general anesthesia because of comorbidities
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Complete enteroscopy rates | up to one year
  Definition of total visualization of small bowel: cecum was reached via antegrade route or antrum was reached via retrograde route; submucosal india ink was observed form 2rd SBE.

SECONDARY OUTCOMES:
Oral insertion depth | up to one year
  Depth of maximal insertion is measured as follow:
  1. Counting folds on withdrawal---fold-counting method;
  2. shorten scope on Treitz ligation and deepest site.
Diagnostic yield | up to one year
  Inflammatory changes Ulcer Angiodysplasia Tumor Diverticulum Others
Procedural time | up to one year
  1. Antegrade insertion time:
     From mouth to Treitz ligation From Treitz ligation to deepest point
  2. Retrograde insertion time:
  From anus to cecum From cecum to marked or deepest site
Adverse events | up to one year
  Pancreatitis Perforation Bleeding Aspiration pneumonia Post-procedural pain score accessed by 100-mm VAS (1h, 3h, 6h, 24h) Others

CONTACTS AND LOCATIONS:
Overall Officials: Shuhui Liang, M.D., Principal Investigator — Associated professor
Locations (2):
- China (2):
  - Endoscopy Center of Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Xijing hospital of Digestive Diseases, Xi'an, Shaanxi